CLINICAL TRIAL: NCT00255294
Title: Non-Comparative Contraceptive Effectiveness Trial of Cellulose Sulfate (CS) Gel
Brief Title: Contraceptive Effectiveness Trial of Cellulose Sulfate Gel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CONRAD (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C02-085
Record Dates: First submitted 2005-11-17; First posted 2005-11-18 (Estimated); Last update posted 2005-11-18 (Estimated); Status verified 2005-11

CONDITIONS: Contraception

INTERVENTIONS:
Drug: Cellulose sulfate vaginal gel

SUMMARY:
This study will evaluate the contraceptive effectiveness of cellulose sulfate vaginal gel in preventing pregnancy when used for 6 months.

DETAILED DESCRIPTION:
Cellulose sulfate has been shown in preclinical studies to have both contraceptive and antimicrobial properties. Clinical safety studies have shown it to be safe for use up to six days in women and 7 days in men, and ongoing studies are assessing its safety for twice daily use for 14 days in women. This study will evaluate its contraceptive effectiveness in women who use it for 6 months.

ELIGIBILITY:
Both partners:

1. Have undergone informed consent procedures as outlined in Section VIII.B.1.
2. In a stable, mutually monogamous relationship for at least three months and anticipating no change in the next 30 weeks.
3. Willing to have coital frequency of at least four times per month on average while in the study.
4. Not actively desiring pregnancy and are willing to accept an unknown risk of pregnancy for the next 30 weeks.
5. Planning to reside in area for 30 weeks after enrollment.
6. Agree to use the study product as instructed at each act of intercourse during the next 30 weeks and to use no other method of contraception (Except: 1) ECPs when indicated, see Section VIII.C.5, or, 2) a barrier method (e.g. Gynol II, condoms) from pre-enrollment until the start of the first post-enrollment menses, see Section VIII.B.4).
7. Willing and able to comply with study procedures.
8. Do not have a known sensitivity or allergy to any vaginal preparations containing glycerin, sorbitol, carbomer, or benzyl alcohol. (Gyne-Lotrimin cream and Cleocin cream contain benzyl alcohol. Replens and Metrogel contain carbomer. K-Y jelly and Replens contain glycerin.)
9. Not known or suspected to be infected by HIV and are at low risk for HIV and other STIs, by virtue of:

   1. Only one sexual partner in the past six months
   2. Not diagnosed with or treated for any STI in the past six months. Note: Individuals with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be enrolled.
   3. Have not shared injection drug needles within the past six months
   4. Do not have any other risk factors known to the clinician or site staff
10. Do not have any other conditions that, in the opinion of the investigator or clinician, would constitute contraindications to participation in the study, would complicate interpretation of data from the participant, or would compromise the participant's ability to comply with the study protocol, such as any major chronic illness including cancer, serious autoimmune disease, substance abuse or a major psychiatric disorder (e.g. schizophrenia).
11. Have not participated in any other investigational trial within 30 days prior to enrollment and have not previously participated in this or any other study involving CS.

Female partner only:

1. Between 18 and 40 years of age, inclusive.
2. Negative pregnancy test at pre-enrollment and enrollment.
3. Regular menstrual cycles (every 21-35 days) for the last two cycles, by participant report.
4. If recently pregnant, must be at least six weeks since the end of the last pregnancy. Must have had two spontaneous menses since the resolution of the last pregnancy.
5. If recently used hormonal contraception:

   1. Combined progestin/estrogen contraceptives (oral/injectable/patch/ring) and progestin-only implant: Must have experienced the withdrawal bleed at the end of the last cycle of use and one subsequent spontaneous menses 21-35 days later.
   2. Progestin-only injectables: Must be at least ten months after the last injection, with two spontaneous menses 21-35 days apart after the last injection.
   3. EC: must have had at least one menses following EC use.
6. No history suggestive of infertility. Infertility is defined as any of the following:

   1. Known history of a fertility problem or sterilization.
   2. Previous ectopic pregnancy or hospitalization for pelvic infection (PID), unless participant has had a spontaneous (without assisted reproductive technology procedures) intrauterine pregnancy afterwards.
   3. Previous pelvic surgery if participant was told that the surgery may lead to a fertility problem or when the PI feels it may have affected fertility.
   4. Abnormalities on pelvic examination at enrollment that may impair fertility (e.g. large fibroids, adnexal masses)
   5. Known history of endometriosis, documented by laparoscopy or laparotomy.
7. Not currently breastfeeding.
8. No Trichomonas on wet prep.
9. No absolute medical contraindication to pregnancy.
10. No vaginal or cervical anatomic abnormality identified by examination and precluding proper placement or retention of the study product.
11. Willing to return to the clinic for scheduled follow-up visits.

Male partner only:

1. At least 18 years of age.
2. No known history of infertility or vasectomy.
3. Has not had sex with a man in the last six months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200
Dates: Start 2005-01; Study Completion 2005-10

PRIMARY OUTCOMES:
1. To estimate the cumulative probability of pregnancy for six months and six cycles of typical use of the CS gel.
2. To estimate the cumulative probability of pregnancy for six cycles of consistent use of the CS gel.
3. To estimate the cumulative probability of study discontinuation through six months of CS gel use.

SECONDARY OUTCOMES:
1. To assess the acceptability of CS gel among female and male users
2. To assess the consistency of use of CS gel among study participants
3. To estimate the frequency of abnormal cytology, candidiasis, urinary tract infections, bacterial vaginosis, and genital irritation during six months of CS gel use.
4. To identify any serious adverse events or patterns of unanticipated adverse events related to the use of CS gel.

CONTACTS AND LOCATIONS:
Overall Officials: Christine K Mauck, MD, Study Director — CONRAD
Locations (1):
- California Family Health Council, Los Angeles, California, United States